CLINICAL TRIAL: NCT05963698
Title: The Fourth Left Atrial Appendage Occlusion Study (LAAOS-4)
Brief Title: The Fourth Left Atrial Appendage Occlusion Study
Acronym: LAAOS-4
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: McMaster University (Other); Population Health Research Institute (Other); Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LAAOS-4
Record Dates: First submitted 2023-07-05; First posted 2023-07-27 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-09

CONDITIONS: Atrial Fibrillation; Stroke, Ischemic; Systemic Embolism
Keywords: WATCHMAN; Left Atrial Appendage (LAA); LAA Device; Left Atrial Appendage Occlusion
MeSH Terms: conditions — Atrial Fibrillation; Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Outcomes Assessor
Masking Description: Events Adjudication Committee is blinded to intervention assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- WATCHMAN device (Experimental): Participants will undergo endovascular left atrial appendage occlusion with the WATCHMAN device
  Interventions: Device: WATCHMAN device
- Standard Care (No Intervention): Participants will receive local, standard medical care

INTERVENTIONS:
Device: WATCHMAN device — Participants will undergo endovascular left atrial appendage occlusion with the WATCHMAN device
  Arms: WATCHMAN device

SUMMARY:
LAAOS-4 aims to determine if catheter-based endovascular left atrial appendage occlusion prevents ischemic stroke or systemic embolism in participants with atrial fibrillation, who remain at high risk of stroke, despite receiving ongoing treatment with oral anticoagulation.

DETAILED DESCRIPTION:
LAAOS-4 is a multicentre, prospective, open-label, randomized controlled trial with blinded assessment of endpoints (PROBE) to determine if catheter-based endovascular left atrial appendage occlusion prevents ischemic stroke or systemic embolism in participants with atrial fibrillation, who remain at high risk of stroke, despite receiving ongoing treatment with oral anticoagulation.

ELIGIBILITY:
Inclusion Criteria:

1. (a) Persistent or permanent atrial fibrillation OR (b) Paroxysmal atrial fibrillation in participants with a history of ischemic stroke or systemic embolism
2. Increased risk of stroke, defined as a CHA2DS2-VASc stroke risk score of ≥ 4. [Note: the acronym CHA2DS2-VASc stands for congestive heart failure, hypertension, age ≥75 (doubled), diabetes, stroke (doubled), vascular disease, age 65 to 74 and sex category (female).]
3. Treatment with oral anticoagulants (Vitamin K agonist or factor Xa inhibitor) for at least 90 days prior to enrollment, AND no documented plan to discontinue treatment with oral anticoagulants for the expected duration of the trial.

Exclusion Criteria:

1. Age < 18 years
2. Current left atrial appendage thrombus
3. Prior left atrial appendage occlusion or removal (surgical or percutaneous)
4. Prior percutaneous atrial septal defect or patent foramen ovale closure
5. Prior atrial fibrillation ablation unless evidence of recurrent qualifying atrial fibrillation present at least 30 days following ablation
6. Planned atrial fibrillation ablation within 90 days of enrollment
7. Individuals being treated with direct thrombin inhibitors
8. Women of childbearing potential unless they agree to employ effective birth control methods throughout the study
9. Anticipated life-expectancy of < 2 years
10. Patient unable or willing to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2029-09-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Ischemic stroke or systemic embolism | The study duration is event-driven. The primary analysis will be performed through study completion, once 265 primary efficacy endpoint events have occurred (an estimated average follow-up of 4 years).
  The primary efficacy variable is the time from randomization to first occurrence of any of the components of the composite outcome (adjudicated) over the duration of follow-up, including:
  * Ischemic stroke (Strokes of undetermined etiology will be treated as ischemic stroke)
  * Systemic embolism

SECONDARY OUTCOMES:
All-cause stroke or systemic embolism | Will be evaluated once primary outcome meets statistical significance. The primary analysis will be performed through study completion, once 265 primary efficacy endpoint events have occurred (an estimated average follow-up of 4 years).
  Secondary efficacy outcomes will be evaluated in a hierarchical fashion only when the primary outcome meets statistical significance in the specified order:
  Time from randomization to first occurrence of all-cause stroke or systemic embolism
All-cause stroke, systemic embolism, or transient ischemic attack (TIA) | Will be evaluated once primary outcome meets statistical significance. The primary analysis will be performed through study completion, once 265 primary efficacy endpoint events have occurred (an estimated average follow-up of 4 years).
  Time from randomization to first occurrence of all-cause stroke, systemic embolism or transient ischemic attack (TIA)
Montreal Cognitive Assessment (MoCA) Score | Will be evaluated once primary outcome meets statistical significance. The primary analysis will be performed through study completion, once 265 primary efficacy endpoint events have occurred (an estimated average follow-up of 4 years).
  Proportion of participants with a decrease of two or more points on the MoCA score at either year 2 or end of study
New disabling ischemic strokes | Will be evaluated once primary outcome meets statistical significance. The primary analysis will be performed through study completion, once 265 primary efficacy endpoint events have occurred (an estimated average follow-up of 4 years).
  Time from randomization to first occurrence of disabling ischemic strokes with modified Rankin Score (mRS) >2, measured at 90 days post-stroke
Cardiovascular mortality | Will be evaluated once primary outcome meets statistical significance. The primary analysis will be performed through study completion, once 265 primary efficacy endpoint events have occurred (an estimated average follow-up of 4 years).
  Time from randomization to cardiovascular mortality
All-cause mortality | Will be evaluated once primary outcome meets statistical significance. The primary analysis will be performed through study completion, once 265 primary efficacy endpoint events have occurred (an estimated average follow-up of 4 years).
  Time from randomization to all-cause mortality

OTHER OUTCOMES:
Non-procedural Major Bleeding | Will be evaluated once primary outcome meets statistical significance. The primary analysis will be performed through study completion, once 265 primary efficacy endpoint events have occurred (an estimated average follow-up of 4 years).
  Proportion of participants with non-procedural Major Bleeding (International Society on Thrombosis and Haemostasis (ISTH) definition; excluding WATCHMAN-related bleeding within 14 days of implant)
Hospitalization for any cause | Will be evaluated once primary outcome meets statistical significance. The primary analysis will be performed through study completion, once 265 primary efficacy endpoint events have occurred (an estimated average follow-up of 4 years).
  Time from randomization to first occurrence of hospitalization for any cause
Heart failure hospitalization or emergency department/clinic visit for intensification of heart failure related therapy | Will be evaluated once primary outcome meets statistical significance. The primary analysis will be performed through study completion, once 265 primary efficacy endpoint events have occurred (an estimated average follow-up of 4 years).
  Time from randomization to first occurrence of heart failure hospitalization or emergency department/clinic visit for intensification of heart failure related therapy
Myocardial Infarction | Will be evaluated once primary outcome meets statistical significance. The primary analysis will be performed through study completion, once 265 primary efficacy endpoint events have occurred (an estimated average follow-up of 4 years).
  Time from randomization to first occurrence of Myocardial Infarction (4th Universal definition)
Device and procedural-related outcomes: Device-related thrombus | Will be evaluated once primary outcome meets statistical significance. The primary analysis will be performed through study completion, once 265 primary efficacy endpoint events have occurred (an estimated average follow-up of 4 years).
  Proportion of participants with device-related thrombus (thrombus formed on the surface of the WATCHMAN device)
Device and procedural-related outcomes: Incomplete left atrial appendage (LAA) closure | Will be evaluated once primary outcome meets statistical significance. The primary analysis will be performed through study completion, once 265 primary efficacy endpoint events have occurred (an estimated average follow-up of 4 years).
  Proportion of participants with incomplete LAA closure
Device and procedural-related outcomes: Peri-procedural major bleeding | Will be evaluated once primary outcome meets statistical significance. The primary analysis will be performed through study completion, once 265 primary efficacy endpoint events have occurred (an estimated average follow-up of 4 years).
  Proportion of participants with peri-procedural major bleeding (ISTH definition; within 14 days following the procedure)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Healey, Principal Investigator — Hamilton Health Sciences Corporation
Locations (106):
- United States (41):
  - Affinity Hospital dba Grandview Medical Center, Birmingham, Alabama
  - Arrhythmia Research Group, Jonesboro, Arkansas
  - Memorial Health Services, Fountain Valley, California
  - Loma Linda University Health, Loma Linda, California
  - Sutter Valley Hospitals dba Sutter Institute for Medical Research, Sacramento, California
  - St. Vincent's Health System, Jacksonville, Florida
  - The University of South Florida, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - St Luke's Regional Medical Center, Ltd, Boise, Idaho
  - Kootenai Health Inc., Coeur d'Alene, Idaho
  - Northwestern University, Evanston, Illinois
  - Cardiovascular Medicine, PLLC and Unity Point Trinity Rock Island, Rock Island, Illinois
  - Community Health Network Inc., Indianapolis, Indiana
  - MercyOne Iowa Heart Center, West Des Moines, Iowa
  - University of Kansas Medical Center Research Institute, Inc., Kansas City, Kansas
  - Babtist Health Lexington, Lexington, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - University of Maryland Baltimore, Baltimore, Maryland
  - Lahey Clinic Inc., Burlington, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - The Feinstein Institutes for Medical Research, Manhasset, New York
  - Cornell University for and on behalf of its Joan & Sanford I. Weill Medical College and The New York Presbyterian Hospital, New York, New York
  - NYU Grossman School of Medicine, New York, New York
  - Mission Hospital HCA, Asheville, North Carolina
  - Aultman Hospital, Canton, Ohio
  - TriHealth Inc., Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Pennsylvania State University and The Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - The Trustees of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center (UPMC) Presbyterian Heart and Vascular Institute, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Glanecare, Inc. d/b/a HCA Florida Brandon Hospital, Brentwood, Tennessee
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
  - Baylor Research Institute, Dallas, Texas
  - Heart Rhythm Associates, The Woodlands, Texas
  - CHRISTUS Northeast Texas Health System, Tyler, Texas
  - The Rector and Visitors of the University of Virginia, Charlottesville, Virginia
  - CommonSpirit Health Research Institute, Tacoma, Washington
  - The Medical College of Wisconsin, Milwaukee, Wisconsin
- Belgium (7):
  - Imeldaziekenhuis, Bonheiden, Antwerpen
  - AZORG vzw and Hartcentrum Aalst, Aalst, East-Flanders
  - ASBL CHU Helora - Hôpital de La Louvière - site Jolimont, La Louvière, Hainaut
  - CHR de la Citadelle, Liège, Liège
  - AZ Glorieux, Ronse, Oost-Vlaanderen
  - AZ Delta VZW, Roeselare, West-Vlaanderen
  - Universitair Ziekenhuis Brussel, Brussels
- Canada (23):
  - University of Calgary, Calgary, Alberta
  - Vancouver Coastal Health Authority, Vancouver, British Columbia
  - St. Boniface Hospital Inc., Winnipeg, Manitoba
  - Circulate Cardiac & Vascular Centre (CCVC), Burlington, Ontario
  - Cambridge Cardiac Care Inc., Cambridge, Ontario
  - Hamilton Health Sciences Corp, Hamilton, Ontario
  - Research St. Joseph's - Hamilton, Hamilton, Ontario
  - Waterloo Wellington Cardiovascular Research Institute (WWCRI), Kitchener, Ontario
  - Lawson Health Research Institute, London, Ontario
  - Southlake Regional Health Centre, Newmarket, Ontario
  - Partners in Advanced Cardiac Evaluation (PACE), Newmarket, Ontario
  - Ottawa Heart Institute Research Corp, Ottawa, Ontario
  - Niagara Health System - Niagara Falls, St. Catharines, Ontario
  - Niagara Health Systems - St. Catharines, St. Catharines, Ontario
  - Sunnybrook Health Sciences Center, Toronto, Ontario
  - Lawrence Park Cardiology, Toronto, Ontario
  - Unity Health Toronto, Toronto, Ontario
  - Institut de Cardiologie de Montreal (ICM), Montreal, Quebec
  - Centre hospitalier de l'Université de Montréal, Montreal, Quebec
  - Institut universitaire de cardiologie et de pneumologie de Québec-Université Laval, Québec, Quebec
  - Centre intégré universitaire de santé et de services sociaux de l'Estrie - Centre hospitalier universitaire de Sherbrooke (CIUSSS de l'Estrie - CHUS), Sherbrooke, Quebec
  - Prairie Valscular Research Inc. (PVRI), Regina, Saskatchewan
  - Saskatchewan Health Authority, Saskatoon, Saskatchewan
- Denmark (5):
  - Region Hospital Viborg, Viborg, Central Jutland
  - Aarhus University Hospital (AUH), Aarhus, Region Midt
  - Esbjerg & Grindsted Hospital - University Hospital of Southern Denmark, Esbjerg, Region Syddanmark
  - North Denmark Regional Hospital, Hjørring
  - Odense Universitets Hospital, Odense C
- France (5):
  - Infirmerie Protestante de Lyon, Caluire-et-Cuire, Auvergne-Rhône-Alpes
  - Clinique Pasteur, Toulouse, Occitanie
  - Hôpital Bichat, Paris
  - European Georges Pompidou Hospital, Paris
  - Centre Cardiologique due Nord, Saint-Denis
- Germany (14):
  - Städtisches Klinikum Karsruhe gGmbH, Karlsruhe, Baden-Wurttemberg
  - CVC Rhein-Main GmbH, Frankfurt am Main, Hesse
  - MVZ CCB Frankfurt und Main-Taunus GbR, Frankfurt am Main, Hesse
  - Johann Wolfgang Goethe Universität Franfurt - Universitätsklinikum Franfurt, Frankfurt am Main, Hesse
  - Krankenhausbetriebsgesellschaft Bad Oeynhausen mbH, Bad Oeynhausen, North Rhine-Westphalia
  - Westpfalz-Klinikum GmbH, Kaiserslautern, Rhineland-Palatinate
  - Herzzentrum Leipzig GmbH, Leipzig, Saxony
  - Universitätsklinikum Schleswig - Holstein, Lübeck, Schleswig-Holstein
  - Katholisches Krankenhaus "St. Johann Nepomuk", Erfurt, Thuringia
  - Charité Universitätsmedizin Berlin, Berlin
  - Charité - Universitätsmedizin Berlin, Berlin
  - Asklepios Kliniken Hamburg GmbH, Hamburg
  - Universitätsklinikum Hamburg-Eppendorf (UKE), Hamburg
  - Universitätsklinikum Heidelberg, Heidelberg
- Fondazione Poliambulanza Istituto Ospedaliero, Brescia, Italy
- American Heart of Poland SA, Ustroń, Poland
- Spain (4):
  - Hospital Álvaro Cunqueiro, Vigo, Pontevedra
  - Complejo Asistencial Universitario de León, León
  - Universitario La Luz - Grupo Quirónsalud, Madrid
  - Hospital Clínico Universitario de Valladolid, Valladolid
- United Kingdom (5):
  - University Hospitals of Leicester NHS Trust, Leicester, Leicestershire
  - Oxford University Hospitals NHS Foundation Trust, Oxford, Oxfordshire
  - University Hospitals Coventry and Warwickshire, Coventry, West Midlands
  - University Hospitals Sussex NHS Trust, Worthing, West Sussex
  - Liverpool Heart and Chest Hospital NHS Foundation Trust, Liverpool

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grifoni E, Pagni B, Sansone T, Baldini M, Bertini E, Giannoni S, Di Donato I, Sivieri I, Iandoli G, Mannini M, Giglio E, Vescera V, Brai E, Signorini I, Cosentino E, Micheletti I, Cioni E, Pelagalli G, Dei A, Giordano A, Dainelli F, Romagnoli M, Mattaliano C, Schipani E, Murgida GS, Di Martino S, Francolini V, Masotti L. Clinical Features, Management, and Recurrence of Acute Ischemic Stroke Occurring in Patients on Oral Anticoagulant Treatment for Nonvalvular Atrial Fibrillation: A Real-World Retrospective Study. Neurologist. 2024 Nov 1;29(6):329-338. doi: 10.1097/NRL.0000000000000579. PMID 39344366